CLINICAL TRIAL: NCT00257335
Title: A Phase II Protocol of Intensity-Modulated Radiotherapy for Treatment of Previously Irradiated Recurrent Head and Neck Cancer
Brief Title: Intensity-Modulated Radiotherapy for Recurrent Head and Neck Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to no patient enrollment this study was withdrawn/closed
Sponsor: Nilam Ramsinghani (Other)
Responsible Party: Sponsor-Investigator, Nilam Ramsinghani, Dr. Nilam Ramsinghani, University of California, Irvine
Organization: University of California, Irvine (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCI 03-58
Record Dates: First submitted 2005-11-21; First posted 2005-11-22 (Estimated); Last update posted 2017-07-31 (Actual); Status verified 2017-07

CONDITIONS: Carcinoma of the Head and Neck
Keywords: Carcinoma of the head and neck

INTERVENTIONS:
Procedure: IMRT

SUMMARY:
To demonstrate safety and efficacy of intensity-modulated radiotherapy (IMRT) for treatment of previously irradiated recurrent head and neck cancer.

Specific Aims: Identify acute and late toxicities, response rates, locoregional control, disease free survival, and overall survival with IMRT. Also, tumor response, the amount of tumor shrinkage or reduction, will be analyzed.

Rationale: Recurrent head and neck cancer is regarded as having limited treatment modalities since salvage surgery can only be accomplished on limited subgroups of patients. Chemotherapy has not shown clear clinical benefits and has significant toxicity. Re-irradiation has been used as a treatment modality. However, the re-irradiation dose is limited by significant toxicity that occurs with the cumulative dose of radiation. The use of IMRT can give a high dose to the recurrent tumor while limiting the dose to critical structures in the vicinity of the reirradiated volume thereby limiting toxicity and treating the recurrence to an adequate dose.

The number of subjects was determined from 2 stage design with a historical control group as comparison, and these numbers of subjects were found to be 40.

It is assumed that this treatment regimen will not be of further interest if the true response rate is less than 32.6% (Po0.326). It is also assumed that a true response rate of 53% or more (P10.53) would be of considerable interest in the treatment of recurrent head and neck cancer. The type I error (the probability of rejecting the hypothesis that the proportion responding to the treatment is less than or equal to Po when this hypothesis is actually true) is 0.05.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have pathologically confirmed recurrence (reappearance of previously cleared) of a squamous cell cancer primary located in the upper aerodigestive tract or a second squamous cell primary. Patients may have experienced more than one recurrence as long as the first recurrence occurred greater than 6 months following the end of the prior RT. Pathology slides from primary as well as recurrence must to be obtained for review by UCI Department of Pathology to confirm histology and patient eligibility. Previous radiation records including simulation and portal films must be submitted to the UCI Department of Radiation Oncology for review of treated areas and to assure that spinal cord tolerance is not exceeded.
2. The recurrence or second primary must have defined bidimensional measurement as follows: All tumor measurements must be recorded in centimeters and should consist of the two longest perpendicular cross-diameters. Patients will be separately assessed for response by physical exam and by CT scan with contrast (unless contraindicated) or MRI scan with T1 contrast with gadolinium (unless contraindicated) and T2 sequences prior to and two months following completion of therapy. Both the clinical (physical exam) and radiographic (CT or MRI) response will be recorded on the study forms.
3. Recurrence or second primary must be confined to the head and neck above the clavicle.
4. The patient must not be a candidate for or refuses complete surgical (re)resection.
5. The majority (>75%) of the tumor volume must have been in areas previously irradiated to >45 Gy. The previous irradiation must not exceed a maximum of 75 Gy.
6. Primary and recurrent cancer treatment cumulative radiation dose must limit total spinal cord dose to 50 Gy.
7. Patients must be at least 1 month from prior chemotherapy and radiation therapy.
8. Karnofsky status 60 or greater. (appendix)
9. WBC >4000/mm3, granulocytes >2,000/mm3, platelets >100,000/mm3, serum bilirubin <1.5 mg/dl, creatinine <1.8 mg/dl within one month from enrollment in protocol.
10. If liver chemistries are above normal limits, a liver ultrasound or CT will be required.
11. Patient must not have a history of other invasive malignancies within the past five years, excluding non-melanomatous skin cancer or cervical cancer in-situ.

Exclusion Criteria

1. Distant metastases.
2. History of other invasive malignancies within the past five years excluding non-melanomatous skin cancer or cervical cancer in-situ.
3. Medical condition, which would impede patient tolerance of therapy, completion of therapy or limit survival.
4. Women who are pregnant will be excluded from this trial. A pregnancy test will be offered to women of child bearing age who are otherwise eligible for the protocol.
5. Patients under 18 years of age will be excluded since head and neck cancer is unlikely and due to risk of long term toxicity from radiation including secondary malignancy
6. Patients on any treatment currently for the recurrent head and neck cancer
7. Patients have any untreated infection
8. Patients are candidate for complete surgical resection.
9. Patients have the previous irradiation exceeded a maximum of 75 Gy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2004-10-14; Primary Completion 2007-06-12 (Actual); Study Completion 2007-06-12 (Actual)

PRIMARY OUTCOMES:
Identify acute and late toxicities and response rates

CONTACTS AND LOCATIONS:
Overall Officials: Nilam Ramshinghani, MD, Principal Investigator — Chao Family Comprehensive Cancer Center